CLINICAL TRIAL: NCT02966457
Title: A Randomized Clinical Study of the Decolonization of MDR Gram-negative Bacteria in Patients With Haematological Malignancies
Brief Title: A Study of DEcolonization in Patients With HAematological Malignancies (DEHAM)
Acronym: DEHAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Minsk Scientific-Practical Center for Surgery, Transplantation and Hematology (Other Government)
Collaborators: Belarusian State Medical University (Other)
Responsible Party: Principal Investigator, Ihar Iskrou, Head of Cell Transplant Division, Minsk Scientific-Practical Center for Surgery, Transplantation and Hematology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HEM-3_1
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Hematological Infection
Keywords: hematological infection, decolonization
MeSH Terms: interventions — colistinmethanesulfonic acid; Colistin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Selective intestinal decolonization (Experimental): Drug: Decolonization with Colistimethate sodium (2 mln I.U. 4x/day PO) for 14 days
  Interventions: Drug: Colistimethate Sodium
- "Wait and watch" strategy (No Intervention): Group without decolonization interventions

INTERVENTIONS:
Drug: Colistimethate Sodium — Selective oral intestinal decolonization
  Other Names: Colistin
  Arms: Selective intestinal decolonization

SUMMARY:
MDR (multidrug resistant) gram-negative bacteria have emerged as an important cause of bloodstream infection in hospitalized patients, especially in immunocompromised hosts. It was previously shown, that intestinal colonization with extended-spectrum β-lactamases (ESBL)-producing or carbapenem-resistant Enterobacteriaceae, carbapenem-resistant A. baumannii and P. aeruginosa) is a clinical predictor of bloodstream infections in patients with haematological malignancies and/or haematopoietic stem cell transplantation [Stoma I. et al., 2016].

To the investigators knowledge no randomized, placebo-controlled clinical trial has been performed to study the efficacy and safety of selective intestinal decolonization strategies in high-risk patients with haematological malignancies. Possible decolonization of MDR gram-negative bacteria in haematological patients could be important for the patient by reducing the risk of infection and for the community by reducing the risk of transmission.

The purpose of the proposed study is to assess the efficacy and safety of selective intestinal decolonization of MDR gram-negative bacteria with oral administration of Colistimethate sodium in high risk patients with haematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Microbiologically proven rectal carriage of ESBL-producing Enterobacteriaceae or carbapenem-resistant Enterobacteriaceae, A. baumannii, P. aeruginosa without signs and symptoms of active infection.
2. Patient must give written informed consent to participate in the study. The informed consent can be given by the legal representative if necessary.

Exclusion Criteria:

1. Active bacterial, viral, fungal or protozoal infection
2. Women who are pregnant or nursing
3. Antibacterial therapy in previous 10 days
4. Contraindication to the use of one of the study drugs (including known hypersensitivity)
5. Patient already enrolled in another study, or in the present study for a previous episode
6. Psychiatric disorder or unable to understand or to follow the protocol directions
7. Resistance of the primarily isolated colonizing microorganism to polymyxin antibiotics proven by methods of polymerase chain reaction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Rate of eradication of ESBL-producing or carbapenem-resistant Enterobacteriaceae, carbapenem-resistant A. baumannii or P. aeruginosa at day 21 post-treatment | 21 days

SECONDARY OUTCOMES:
Rate of resistance of isolated on day 21 post-treatment Enterobacteriaceae, A. baumannii, P. aeruginosa to polymyxin antibiotics | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Ihar Iskrou, Ph.D., Study Chair — Republican Center of Hematology and Bone Marrow Transplantation
Locations (1):
- Republican Center of Hematology and Bone Marrow Transplantation, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stoma I, Karpov I, Milanovich N, Uss A, Iskrov I. Risk factors for mortality in patients with bloodstream infections during the pre-engraftment period after hematopoietic stem cell transplantation. Blood Res. 2016 Jun;51(2):102-6. doi: 10.5045/br.2016.51.2.102. Epub 2016 Jun 23. PMID 27382554
- [Background] Rieg S, Kupper MF, de With K, Serr A, Bohnert JA, Kern WV. Intestinal decolonization of Enterobacteriaceae producing extended-spectrum beta-lactamases (ESBL): a retrospective observational study in patients at risk for infection and a brief review of the literature. BMC Infect Dis. 2015 Oct 28;15:475. doi: 10.1186/s12879-015-1225-0. PMID 26511929
- [Derived] Stoma I, Karpov I, Iskrov I, Krivenko S, Uss A, Vlasenkova S, Lendina I, Cherniak V, Suvorov D. Decolonization of Intestinal Carriage of MDR/XDR Gram-Negative Bacteria with Oral Colistin in Patients with Hematological Malignancies: Results of a Randomized Controlled Trial. Mediterr J Hematol Infect Dis. 2018 May 1;10(1):e2018030. doi: 10.4084/MJHID.2018.030. eCollection 2018. PMID 29755707